CLINICAL TRIAL: NCT02929602
Title: PRL0706: Analgesic Use and Effectiveness
Brief Title: Analgesic Use and Effectiveness for Dental Procedures
Status: Completed | Type: Observational
Sponsor: Pearl Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRL0706; U01DE016755 (NIH)
Record Dates: First submitted 2016-02-05; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: prescribing; effectiveness; dental; opioid; analgesic
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Opioid analgesics prescribed by dentists may contribute to the larger national issue of the use and abuse of the drug. On occasion dental pain may be sufficiently severe to support the use of opioids. This study used both dentist and patient input to evaluate the use of opioid and over-the-counter analgesics following one of seven coded common dental procedures. The study includes a five day patient follow up assessment of the effectiveness of the analgesic. Baseline questionnaires were completed by eligible participants, and they responded to the day 5 follow up questionnaires.

DETAILED DESCRIPTION:
Specific Aims The overall objective of the proposed study is to determine (1) the pattern of analgesic prescriptions (Rx and OTC) and recommendations (OTC) in dental practices; and (2) the effectiveness of and side effects associated with these medications as measured by patientreported outcomes (PROs).

Specific Aim 1: To document (a) dentists' postprocedural prescriptions and recommendations for analgesic medication: and (b) the effectiveness of these medications and side effects associated with their use as measured by PROs.

Specific Aim 2: To analyze by procedure class and anticipated pain severity the PROs of Rx and OTC analgesic medications.

Specific Aim 3: Determine the incidence of analgesic side effects of Rx and OTC analgesic medications.

The outcomes of Specific Aims 1-3 will be:

* The distribution of dentists' Rx/OTC prescriptions/recommendations by dentists for anticipated pain severity.
* The effectiveness of different types of Rx and OTC analgesics (e.g., Rx NSAIDs vs. OTC NSAIDs, Rx NSAIDs vs. Rx narcotics) by procedure class and anticipated pain severity.
* The incidence of analgesic side effects for Rx and OTC analgesics. Analysis of the results and methods of the proposed research will furthermore serve as guidance in designing a randomized PBRN clinical trial comparing the efficacy of and complications associated with two or more analgesics.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of erupted second molar teeth.
2. Scheduled for treatment in one procedure of the following six procedure classes:

   extraction, endodontic therapy, pulp capping, crown preparation, periodontal surgery, abscess treatment
3. Expected by the P-I to experience postoperative pain sufficient to require an analgesic
4. Permanent dentition (erupted 2nd molar teeth)
5. Capacity to judge pain level
6. Ability and willingness to give verbal consent

Exclusion Criteria:

1. Under treatment for medical disorders, including dementia, Parkinson's disease, depression, severe anxiety, or any other medical condition, that, in the opinion of the P-I, would affect the subject's judgment of postoperative pain
2. Current participation in another dental or medical research study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practice-based study. Patients recruited from the practice sites of PEARL Network dentists.
Sampling Method: Non-Probability Sample
Enrollment: 2773 (Actual)
Dates: Start 2007-06; Primary Completion 2011-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Dentist questionnaire | baseline
  dentists' postprocedural prescriptions were recorded by analgesic class: Opioid, NSAID, or other (Descriptive measures)

SECONDARY OUTCOMES:
Dentist questionnaire - anticipated pain by patients using VAS-5 pain scale | 5 days after the dental procedure
  anticipated pain severity using the VAS-5 pain scale (1-5 scale)
Patient questionnaire - OHIP-14 patient reported outcomes quality of life survey (questionnaire). | 5 days after the dental procedure

OTHER OUTCOMES:
Patient questionnaire - side effects of analgesics post dental procedure | 5 days post dental procedure
  (Descriptive methods were used) to determine side effects: Yes/no, describe for Rx and OTC analgesic medications.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Curro, DMD, PhD, Principal Investigator — Pearl Network
Locations (1):
- PEARL Network Sites, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Will send to the NIDCR.

REFERENCES:
- [Derived] Wong YJ, Keenan J, Hudson K, Bryan H, Naftolin F, Thompson VP, Craig RG, Vena D, Collie D, Wu H, Matthews AG, Grill AC, Curro FA. Opioid, NSAID, and OTC Analgesic Medications for Dental Procedures: PEARL Network Findings. Compend Contin Educ Dent. 2016 Nov/Dec;37(10):710-718. PMID 27875056